CLINICAL TRIAL: NCT00349375
Title: A Multicenter, Double-Blind, Randomized, Active Comparator, Forced-Titration Study to Compare the Efficacy and Safety of the Combination of 145 mg Fenofibrate and 20 or 40 mg Simvastatin With 40 mg Simvastatin Monotherapy in Patients With Mixed Dyslipidemia at Risk of Cardiovascular Disease Not Adequately Controlled by 20 mg Simvastatin Alone
Brief Title: Comparison of the Combination of Fenofibrate and 20 mg Simvastatin Versus 40 mg Simvastatin Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Martine Guy, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C LF0242780-01 05 01; 2005-003270-14
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia Combined, efficacy combination fenofibrate simvastatin
MeSH Terms: conditions — Hyperlipidemias | interventions — Fenofibrate; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Fenofibrate/Simvastatin
- 2 (Experimental)
  Interventions: Drug: Fenofibrate/Simvastatin
- 3 (Active Comparator)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Fenofibrate/Simvastatin — Combination of Fenofibrate 145mg and Simvastatin 20mg
  Arms: 1
Drug: Fenofibrate/Simvastatin — Combination of Fenofibrate and Simvastatin 40 mg
  Arms: 2
Drug: Simvastatin — Simvastatin 40 mg
  Arms: 3

SUMMARY:
Mixed or combined hyperlipidemia is a common metabolic disorder characterized by both hypercholesterolemia and hypertriglyceridemia. Statins and fibrates have complementary mechanisms and can be coadministered to patients with mixed hyperlipidemia. The overall objective of the study is to evaluate the efficacy and safety of combining fenofibrate and simvastatin in patients with mixed hyperlipidemia at risk of cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Mixed dyslipidemia

Exclusion Criteria:

* Known hypersensitivity to fenofibrate or simvastatin
* Pregnant or lactating women
* Contra-indication to fenofibrate or simvastatin
* Unstable or severe cardiac disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Actual)
Dates: Start 2005-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to 24 weeks of treatment in Triglycerides | 12 weeks
Percent change from baseline to 24 weeks of treatment in HDL-C | 12 weeks
Percent change from baseline to 24 weeks of treatment in LDL-C | 12 weeks

SECONDARY OUTCOMES:
Percent change from baseline to 24 weeks of treatment in Triglycerides | 24 weeks
Percent change from baseline to 24 weeks of treatment in HDL-C | 24 weeks
Percent change from baseline to 24 weeks of treatment in LDL-C | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (110):
- Czechia (19):
  - Site 008, Brno
  - Site 009, Brno
  - Site 010, Brno
  - Site 015, Hradisk
  - Site 019, Karlovy Vary
  - Site 014, Kladno
  - Site 005, Nymburk
  - Site 012, Olomouc
  - Site 013, Olomouc
  - Site 007, Pilsen
  - Site 018, Pilsen
  - Site 001, Prague
  - Site 002, Prague
  - Site 003, Prague
  - Site 004, Prague
  - Site 016, Příbram
  - Site 017, Příbram
  - Site 011, Slaný
  - Site 006, Tábor
- Denmark (3):
  - Site 201, Copenhagen
  - Site 205, Copenhagen
  - Site 203, Hvidovre
- France (21):
  - Site 302, Bouliac
  - Site 314, Briollay
  - Site 318, Corsept
  - Site 301, Dijon
  - Site 317, La Montagne
  - Site 321, Le Mesnil En Valee
  - Site 316, Loudon
  - Site 308, Mont-de-Marsan
  - Site 312, Mûrs-Erigné
  - Site 310, Nantes
  - Site 304, Niort
  - Site 319, Orvault
  - Site 306, Paris
  - Site 305, Pouilly-en-Auxois
  - Site 307, Rouen
  - Site 311, Rouen
  - Site 303, Saint-Justin
  - Site 315, Thouars
  - Site 309, Vieux-Condé
  - Site 313, Vihiers
  - Site 320, Vue
- Germany (15):
  - Site 109, Deidesheim
  - Site 108, Frankfurt
  - Site 101, Freiburg im Breisgau
  - Site 111, Hamburg
  - Site 103, Hanover
  - Site 104, Ilvesheim
  - Site 110, Kassel
  - Site 106, Mannheim
  - Site 114, München
  - Site 113, Neu-Anspach
  - Site 105, Offenbach
  - Site 107, Offenbach
  - Site 115, Paderborn Kernstadt
  - Site 102, Rodgau
  - Site 112, Wermsdorf
- Hungary (13):
  - Site 406, Békéscsaba
  - Site 401, Budapest
  - Site 411, Budapest
  - Site 412, Budapest
  - Site 405, Debrecen
  - Site 402, Gyöngyös
  - Site 409, Gyula
  - Site 410, Kecskemét
  - Site 404, Miskolc
  - Site 413, Mosonmagyaróvár
  - Site 407, Orosháza
  - Site 408, Szeged
  - Site 403, Szolnok
- Netherlands (14):
  - Site 511, 's-Hertogenbosch
  - Site 508, Breda
  - Site 509, De Bilt
  - Site 502, Eindhoven
  - Site 514, Eindhoven
  - Site 503, Groningen
  - Site 512, Hengelo
  - Site 506, Leiden
  - Site 507, Nijmegen
  - Site 501, Rotterdam
  - Site 513, Tiel
  - Site 510, Utrecht
  - Site 505, Velp
  - Site 504, Zoetermeer
- Poland (10):
  - Site 606, Chrzanów
  - Site 601, Gdansk
  - Site 603, Katowice
  - Site 609, Sopot
  - Site 602, Warsaw
  - Site 607, Warsaw
  - Site 608, Warsaw
  - Site 605, Wroclaw
  - Site 610, Wroclaw
  - Site 604, Zabrze
- Ukraine (15):
  - Site 701, Dnipropetrovsk
  - Site 702, Dnipropetrovsk
  - Site 709, Dnipropetrovsk
  - Site 712, Donetsk
  - Site 703, Kharkiv
  - Site 705, Kharkiv
  - Site 711, Kharkiv
  - Site 704, Kyiv
  - Site 706, Kyiv
  - Site 707, Kyiv
  - Site 708, Kyiv
  - Site 715, Kyiv
  - Site 713, Luhansk
  - Site 714, Odesa
  - Site 710, Zaporizhya